CLINICAL TRIAL: NCT06248138
Title: Factors Related to the Progression of Non-target Coronary Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mei Gao (Other)
Responsible Party: Sponsor-Investigator, Mei Gao, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(155)
Record Dates: First submitted 2024-01-09; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Coronary Stenosis
Keywords: Coronary heart disease; Atherosclerotic progression; Non-target coronary lesion; Quantitative flow ratio
MeSH Terms: conditions — Coronary Stenosis; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Progression: There is at least one major coronary artery (left main artery, left anterior descending artery, left circumflex artery or the right coronary artery) had non-target lesions, and the coronary artery stenosis rate reached the progressive level on follow-up angiography.
- Non-progression: The rate of coronary stenosis of the non-target lesion did not reach progressive levels during the repeat angiography.

SUMMARY:
The goal of this observational study is to learn about correlation between traditional risk factors and emerging risk factors on the progression of non-target coronary lesions in patients with non-target lesions on at least two coronary angiographies at the First Affiliated Hospital of Shandong First Medical University. The main question it aims to answer is what the correlation between emerging risk factors and progression of coronary non-target lesions, and try to explore the powerful predictors of progression of coronary non-target lesions and cardiovascular events.

Participants will be divided into two groups based on coronary angiography results:

1. progress group:There is at least one major coronary artery (left main artery, left anterior descending artery, left circumflex artery or the right coronary artery) had non-target lesions, and the coronary artery stenosis rate reached the progressive level on follow-up angiography.
2. Non-progress groups: On repeat angiography, the rate of coronary stenosis did not reach progressive levels.

DETAILED DESCRIPTION:
The laboratory and auxiliary examination indexes of the study participants were collected prior to two coronary angiography (CAG) procedures, encompassing blood cell counts, glucose metabolism, lipid metabolism, renal function, cardiac function, inflammatory factors, etc. Quantitative flow fraction (QFR) was employed for assigning values to coronary artery images and analyzing lesion information (including plaque progression and non-progression). The correlation between conventional risk factors, lipoprotein(a), homocysteine, and other emerging risk factors with the progression of non-target coronary lesions was analyzed; furthermore, the predictive value of emerging risk factors for non-target coronary lesion progression was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old;
2. Participants underwent at least two coronary angiography examinations in our hospital, and the time interval between the two angiography examinations was ≥12 months;
3. At the first angiography, there is 20% to 70% stenosis in the coronary artery lesion, and no indication or condition for intervention.

Exclusion Criteria:

1. Participants had a documented medical history of various heart diseases, including congenital heart disease, pulmonary heart disease, valvular disease, cardiomyopathy, etc.
2. Angiography or serum collection was conducted within 7 days following the onset of acute myocardial infarction.
3. Exclusion criteria included uncontrolled severe arrhythmia and severe hepatic and renal dysfunction.
4. Patients with tumor or other autoimmune diseases were excluded from the study.
5. Incomplete clinical information, biochemical test information, coronary angiography data, and imaging data were considered as exclusion factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-target lesions who underwent at least two instances of coronary angiography at the First Affiliated Hospital of Shandong First Medical University from January 2017 to present were included in the study.
Sampling Method: Probability Sample
Enrollment: 1111 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between emerging risk factors and progression of coronary non-target lesions. | The estimated period of time over which the event is assessed up to 16 weeks, and from date of grouping until the date of first documented progression whichever came first, assessed up to 60 months.
  To calculate the change of non-target lesion stenosis rate , and get the correlation with homocysteine, lipoprotein(a) and so on by Logistic regression analysis

SECONDARY OUTCOMES:
Association of traditional risk factors and inflammation with the evolution of coronary non-target lesions | The estimated period of time over which the event is assessed up to 16 weeks, and from date of grouping until the date of first documented progression whichever came first, assessed up to 60 months.
  To calculate the change of non-target lesion stenosis rate , and get the correlation with the basic information and inflammation of the participants by Logistic regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: mei Gao, doctor, Study Chair — Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) utilized in this study were obtained from our hospital's healthcare big data cloud platform. In consideration of the data security and privacy protection for study participants, the sharing of this data with other researchers is currently restricted.

REFERENCES:
- [Background] Nakachi T, Kosuge M, Hibi K, Ebina T, Hashiba K, Mitsuhashi T, Endo M, Umemura S, Kimura K. C-reactive protein elevation and rapid angiographic progression of nonculprit lesion in patients with non-ST-segment elevation acute coronary syndrome. Circ J. 2008 Dec;72(12):1953-9. doi: 10.1253/circj.cj-08-0185. Epub 2008 Oct 29. PMID 18957790
- [Background] Xin H, Gong HP, Cai SL, Ning XF, Liu S, Chen ZY, Lian ZX, Zhang R, Zhang QF, Kang WQ, Ge ZM. Elevated lipoprotein-associated phospholipase A2 is associated with progression of nonculprit lesions after percutaneous coronary intervention. Tohoku J Exp Med. 2013 Jun;230(2):97-102. doi: 10.1620/tjem.230.97. PMID 23774398
- [Background] Hartmann M, von Birgelen C, Mintz GS, Stoel MG, Eggebrecht H, Wieneke H, Fahy M, Neumann T, van der Palen J, Louwerenburg HW, Verhorst PM, Erbel R. Relation between lipoprotein(a) and fibrinogen and serial intravascular ultrasound plaque progression in left main coronary arteries. J Am Coll Cardiol. 2006 Aug 1;48(3):446-52. doi: 10.1016/j.jacc.2006.03.047. Epub 2006 Jul 12. PMID 16875967
- [Background] Boroumand MA, Rekabi V, Davoodi G, Amirzadegan A, Saadat S, Abbasi SH, Hamidian R, Poorgholi L. Correlation between lipoprotein(a) serum concentration and severity of coronary artery stenosis in an Iranian population according to Gensini score. Clin Biochem. 2008 Feb;41(3):117-20. doi: 10.1016/j.clinbiochem.2007.10.004. Epub 2007 Oct 16. PMID 17976374
- [Background] Montalescot G, Ankri A, Chadefaux-Vekemans B, Blacher J, Philippe F, Drobinski G, Benzidia R, Kamoun P, Thomas D. Plasma homocysteine and the extent of atherosclerosis in patients with coronary artery disease. Int J Cardiol. 1997 Aug 8;60(3):295-300. doi: 10.1016/s0167-5273(97)00099-5. PMID 9261641
- [Background] Ferraro S, Marano G, Biganzoli EM, Boracchi P, Bongo AS. Prognostic value of cystatin C in acute coronary syndromes: enhancer of atherosclerosis and promising therapeutic target. Clin Chem Lab Med. 2011 Sep;49(9):1397-404. doi: 10.1515/CCLM.2011.607. Epub 2011 May 24. PMID 21605013
- [Result] Authors/Task Force Members; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2019 ESC/EAS guidelines for the management of dyslipidaemias: Lipid modification to reduce cardiovascular risk. Atherosclerosis. 2019 Nov;290:140-205. doi: 10.1016/j.atherosclerosis.2019.08.014. Epub 2019 Aug 31. No abstract available. PMID 31591002
- [Result] Zhang Y, Wu NQ, Li S, Zhu CG, Guo YL, Qing P, Gao Y, Li XL, Liu G, Dong Q, Li JJ. Non-HDL-C is a Better Predictor for the Severity of Coronary Atherosclerosis Compared with LDL-C. Heart Lung Circ. 2016 Oct;25(10):975-81. doi: 10.1016/j.hlc.2016.04.025. PMID 27634241